CLINICAL TRIAL: NCT01762267
Title: Phase 3 Study of Beneficiary Effects of Dietary Approaches to Stop Hypertension (DASH) on the Metabolic Aeffects of Corticosteroids Medications Use
Brief Title: Effects of DASH Diet on Corticosteroids Medication Use
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Isfahan University of Medical Sciences, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DASH in corton therapy
Record Dates: First submitted 2012-12-01; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Nutritional and Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diet intervention, DASH diet (Active Comparator): intervention: nutrition intervention: DASH diet
  Interventions: Other: nutrition intervention
- not intervention, control diet (No Intervention): control weight loss diet

INTERVENTIONS:
Other: nutrition intervention — DASH diet control diet
  Arms: diet intervention, DASH diet

SUMMARY:
To determine the effects of the Dietary Approaches to Stop Hypertension (DASH) diet on the metabolic side effects of corticosteroids medications use.

DETAILED DESCRIPTION:
Objective: To determine the effects of the Dietary Approaches to Stop Hypertension (DASH) diet on the metabolic side effects of corticosteroids medications use.

Design: A randomized clinical trial was undertaken in 60 patients on corticosteroid therapy for 10 weeks. Patients were randomly assigned to a DASH or control diet. Fasting blood sample were measured to determine blood glucose and lipid profile. Blood pressure and anthropometric measurements were measured based on the standard guidelines.

ELIGIBILITY:
Inclusion Criteria:

* patients who were on corticosteroid therapy

Exclusion Criteria:

* refuse to follow the visits

Ages: 27 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
the amount of weight reduction and change of blood pressure | up to 10 weeks
  weight (kg) body mass index (kg/m2) blood pressure (mmHg)

SECONDARY OUTCOMES:
lipid profile, fasting blood glucose | 10 weeks
  measurement of LDL-C (mg/dl), HDL-C (mg/dl), triglyceride (mg/dl), total cholesterol (mg/dl), fasting blood glucose(mg/dl), by the analysis of blood samples and blood pressure(mmHg) and weight (kg), waist circumference (cm), body mass index (kg/m2).

OTHER OUTCOMES:
lipid profile (mg/dl), fasting blood glucose (mg/dl), blood pressure (mmHg), weight reduction (kg) | july

CONTACTS AND LOCATIONS:
Overall Officials: Leila azadbakht, PhD, Study Director — 1. Department of Community Nutrition, School of Nutrition & Food Science, Isfahan University of Medical Science, Isfahan, Iran
Locations (1):
- 1. Department of Community Nutrition, School of Nutrition & Food Science, Isfahan University of Medical Science, Isfahan, Iran